CLINICAL TRIAL: NCT02447406
Title: Phase Ib, Single-arm Study of AZD6094 (Volitinib) in Combination With Docetaxel, in Any Solid Cancer and Sequential Phase II, Single-arm Study of AZD6094 (Volitinib) in Combination With Docetaxel in Advanced Gastric Adenocarcinoma Patients With MET Amplification as a Second Line Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim,PhMD, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-07-169
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD6094 (Volitinib) in combination with docetaxel (Experimental): Phase Ib:Volitinib should be administered at least 200mg orally once a day in 21 days for achieving appropriate antitumor activity.
  Phase II: Subjects will receive Volitinib once daily ( at the MTD determined from Phase Ib) for 21 days as one cycle.
  Docetaxel 60 mg/m2 will be administered via intravenous access once every 3 weeks.
  Interventions: Drug: AZD6094; Drug: docetaxel

INTERVENTIONS:
Drug: AZD6094
  Other Names: Volitinib
Drug: docetaxel

SUMMARY:
Phase Ib/II, single-arm study of AZD6094 (Volitinib) in combination with docetaxel, in advanced gastric adenocarcinoma patients with MET amplification as a second-line treatment.

Phase Ib:Investigational product, dosage and mode of administration Volitinib is an orally available, potent, selective, small molecule c-MET inhibitor.

Volitinib should be administered at least 200mg orally once a day in 21 days for achieving appropriate antitumor activity.

Docetaxel 60 mg/m2 will be administered via intravenous access once every 3 weeks Phase II: Investigational product, dosage and mode of administration Volitinib is an orally available, potent, selective, small molecule c-MET inhibitor. Subjects will receive Volitinib once daily ( at the MTD determined from Phase Ib) for 21 days as one cycle.

Docetaxel 60 mg/m2 will be administered via intravenous access once every 3 weeks.

DETAILED DESCRIPTION:
Volitinib is a potent and selective small molecule c-Met kinase inhibitor. Volitinib was found to inhibit c-Met kinase at the enzyme and cell levels with IC50s of 4 nM for both enzyme and Met phosphorylation in the cell. Consistent with its potent enzyme and cell activity, volitinib was found to inhibit cell growth in vitro against tumors with c-Met gene amplification in the absence of HGF stimulation with IC50s generally below 10 nM. It also potently inhibited HGF-stimulated cell proliferation against tumors with c-Met overexpression or carrying a HGF/c-Met autocrine loop.

In a xenograft model Hs746T with c-Met gene amplification, suboptimal doses 0.6 mg/kg volitinib and 3 mg/kg docetaxel induced TGI(expand) of 55.8% and 80.8%, respectively, whereas combination resulted in a TGI by 101.1%, and statistical significance was seen between combination group and either of mono-therapy group. Plasma exposures of volitinib and docetaxel were determined after last dose at the end of study, and there was no significant difference between combination and single agent on exposures of either volitinib or docetaxel. More importantly, combination was well tolerant and no body weight loss was found in the animals. These results suggested that it would be worthwhile to study the combination use of volitinib and docetaxel in clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. For Phase Ib: Have histologically or cytologically confirmed diagnosis of relapsed or refractory locally advanced or metastatic solid tumors for whom no alternative effective standard therapy is available or for whom standard therapy is considered unsuitable or intolerable.

   - Although it is preferred to enroll patients with solid tumors harboring MET amplification, this will not be an enrollment requirement.

   For Phase II: Advanced gastric adenocarcinoma (including GEJ expand and maybe include in list of abbreviations) that has progressed during or after first-line therapy.
   * The 1st line regimen must have contained doublet 5-fluoropyrimidine and platinum based regimen.
   * Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing doublet 5-fluoropyrimidine and platinum-based regimen could be considered as 1st line therapy.
   * Patients with gastric adenocarcinoma harboring MET amplification by MET FISH.
4. Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the 1st line therapy.
5. Provision or availability of biopsy sample for analysis; e.g mandatory pre-treatment biopsy, or available diagnostic biopsy of sufficient quantity/quality
6. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
7. ECOG performance status 0-1.
8. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
9. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

   * Haemoglobin ≥9.0 g/dL (transfusion allowed)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) > 3 x 109/L
   * Platelet count ≥100 x 109/L (transfusion allowed)
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (does not include patients with Glibert's disease)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   * Serum creatinine ≤1.5 x institutional ULN
10. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and follow up visits.
11. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1 for women of childbearing potential.
12. Provision of consent for mandatory biopsy at progression. (fresh frozen will be mandatory if clinically feasible)

Exclusion Criteria:

1. More than one prior chemotherapy regimen (except for adjuvant/neoadjuvant chemotherapy with more than 6 month wash out period) for the treatment of gastric cancer in the advanced setting.
2. Any previous treatment with MET inhibitors
3. Any previous treatment with docetaxel.
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
5. HER2 positive patients (defined by HER2 3+ by immunohistochemistry or HER2 SISH +)
6. Patients unable to swallow orally administered medication.
7. Treatment with any investigational product during the last 28 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
8. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
9. With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
10. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
11. Resting ECG with measurable QTcB > 480 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
12. Patients with cardiac problem as follows: uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) Baseline Left ventricular ejection fraction below the LLN of <55% measured by echocardiography or institution's LLN for MUGA, Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment
13. Female patients who are breast-feeding or child-bearing and Male or female patients of reproductive potential who are not employing an effective method of contraception
14. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
15. Patients currently receiving (or unable to stop use at least 2 weeks) prior to receiving the first dose of AZD6094, medications known to be potent inhibitors of CYP1A2 or CYP3A4, potent inducers of CYP3A4 or CYP3A4 substrates with a narrow therapeutic range.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Hematologic toxicity and non-hematologic toxicity according to NCI-CTCAE version 4.0 | expected average of 24 weeks
  To determine maximal tolerate dose (MTD) of volitinib when given in combination with fixed dose of docetaxel in any solid cancer
Objective response rate (ORR) by RECIST 1.1 | expected average of 24 weeks
  Phase II:To investigate the efficacy of volitinib when given in combination with docetaxel in patients with advanced gastric adenocarcinoma harboring MET amplification

SECONDARY OUTCOMES:
Duration of response | expected average of 24 weeks
Disease control rate | 8 weeks
Overall survival (OS) | expected average of 24 weeks
progression-free survival (PFS) | expected average of 24 weeks
Number of subjects with Adverse Events as a Measure of safety and tolerability | expected average of 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, Korea, Republic of, South Korea